CLINICAL TRIAL: NCT00400647
Title: A 12-week Multicenter, Randomized, Open Study to Evaluate the Effects of Enteric-coated Mycophenolate Sodium (EC-MPS) in Terms of Quality of Life in Patients With Gastrointestinal (GI) Symptoms Treated With MMF (Mycophenolate Mofetil) After Kidney Transplant.
Brief Title: Gastrointestinal and Health-related Quality of Life in Kidney Transplant Patients Treated With Mycophenolate Mofetil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AES06
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Maintenance Kidney Transplant
Keywords: kidney transplant; enteric-coated mycophenolate sodium; quality of life; gastrointestinal symptoms
MeSH Terms: interventions — Mycophenolic Acid

ARMS (2):
- EC MPS (Experimental): Up to 1440mg taken in two doses
  Interventions: Drug: Enteric-coated Mycophenolate sodium (EC-MPS)
- Mycophenolate mofetil (Active Comparator): 250 mg or 500 mg in two equal doses
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)
  Arms: EC MPS
Drug: Mycophenolate mofetil
  Arms: Mycophenolate mofetil

SUMMARY:
This study will assess the quality of life in renal transplant recipients who require a reduced dose of mycophenolate mofetil (MMF) because of gastrointestinal (GI) side effects and will also access the relationship between mycophenolic acid (MPA) dose in those patients receiving enteric-coated mycophenolate sodium formulation(EC-MPS).

Patients will be evaluated at baseline, 2 weeks after study medicine conversion and then again at 12 weeks post-conversion.

ELIGIBILITY:
Inclusion criteria

1. Patients who are recipients of a renal transplant.
2. Patients treated with an immunosuppressive regiment including MMF before recruitment.
3. Patients suffering from GI side effects related to MMF standard doses or patients treated with a reduced MMF dose to control the aforementioned GI side effects.
4. Patients 18 years or older.
5. Patients who have given written informed consent to participate in the study
6. Patients complying with all study requirements including completing questionnaires and attending to the three study visits.

Exclusion criteria

1. Patients with GI symptoms assumed or known not to be caused by MPA therapy (eg. oral bisphosphonate induced, infectious diarrhea)
2. Acute rejection less than 1 week before recruitment.
3. Females of childbearing potential who are pregnant, planning to get pregnant and/or breast feeding or not willing to practice an approved method of birth control.
4. Presence of psychiatric disorder, such as schizophrenia or major depression, in the investigator's opinion, could interfere with study requirements.
5. Patients undergoing surgery due to acute illness or hospitalized.
6. Existence of any medical condition which, in the investigator's opinion based on anamnesis or medical records, could affect study completion, including but not limiting visual problems or cognitive deterioration.
7. Patients currently treated or who have been treated with any other study drug or treatment within 30 days prior to baseline visit.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of the use of EC-MPS on the quality of life of patients requiring MMF dose reduction due to gastrointestinal symptoms | 12 weeks

SECONDARY OUTCOMES:
To determine whether EC-MPS enables the administration of higher doses with good tolerability, compared with standard MMF treatment, in patients with shown susceptibility to undesirable GI effects | 12 weeks
To measure health-related quality of life (HRQOL) through the GI quality of life index (GIQLI) and the psychological general well-being index (PGWB) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Result] Ortega F, Sanchez-Fructuoso A, Cruzado JM, Gomez-Alamillo JC, Alarcon A, Pallardo L, Morales JM, Oliver J, Guinea G; MYVIDA Study Group. Gastrointestinal quality of life improvement of renal transplant recipients converted from mycophenolate mofetil to enteric-coated mycophenolate sodium drugs or agents: mycophenolate mofetil and enteric-coated mycophenolate sodium. Transplantation. 2011 Aug 27;92(4):426-32. doi: 10.1097/TP.0b013e31822527ca. PMID 21760569